CLINICAL TRIAL: NCT05321316
Title: Nectin-4 Specific LMW PET Probe Imaging in Urothelial Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022KT37
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-N188 (Experimental): Imaging cohort All study participants will be allocated to this arm (single-arm study). Study participants will undergo 68Ga-N188 PET/CT scan.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All study participants will undergo one 18F-FDG PET/CT scan.

SUMMARY:
To evaluate the ability of [68Ga]N188 to detect nectin-4 overexpression in patients with urothelial carcinoma, especially in patients with recurrent or advanced bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, male or female;
2. Heart function is normal;
3. Normal heart function;
4. Estimated survival ≥12 weeks;
5. Good follow-up compliance;
6. presence of at least one measurable target lesion according to RECIST1.1 criteria;
7. Women of childbearing age (15-49 years) must have a negative pregnancy test within 7 days before starting the test; Fertile men and women must agree to use effective contraception to prevent pregnancy during the study period and for 3 months after the test;
8. Patients recommended by clinicians to undergo PET/CT examination for tumor diagnostic staging;
9. The subject patients could fully understand and voluntarily participate in the experiment, and signed the informed consent.

Exclusion Criteria:

1. Serious abnormality of liver, kidney and blood;
2. Pregnant patients;
3. Pregnant and lactation women;

3) unable to lie flat for half an hour; 4) Refuse to join the clinical investigator; 5) Suffering from claustrophobia or other mental diseases; 6) Other conditions that researchers deem unsuitable for participating in the experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 2 years
  SUV is a semi-quantitative analysis index to describe the radioactive uptake of lesions, which has certain reference value for differentiating benign and malignant lesions。 The uptake of the tracer （68Ga-N188） in urothelial carcinoma tumor lesions by measuring SUV on PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No